CLINICAL TRIAL: NCT03100123
Title: A Pilot Study Assessing the Feasibility of a Randomized Controlled Trial Evaluating Aspirin Versus Low-molecular-weight Heparin (LMWH) and Aspirin in Women With Antiphospholipid Syndrome and Pregnancy Loss
Brief Title: AntiPhospholipid Syndrome Low-molecular-weight Heparin Pregnancy Loss Evaluation: The Pilot Study
Acronym: APPLE
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Pilot deemed not feasible by Steering Committee due to recruitment rate.
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO 0807
Record Dates: First submitted 2017-02-21; First posted 2017-04-04 (Actual); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Antiphospholipid Syndrome in Pregnancy; Pregnancy Loss
MeSH Terms: interventions — Aspirin; Heparin, Low-Molecular-Weight; Tinzaparin; Dalteparin; Enoxaparin

STUDY DESIGN:
Intervention Model Description: Eligible and consenting subjects will be assigned to one of two study arms. Randomization is stratified by 'high-risk' or 'non-high risk' laboratory criteria and the timing of pregnancy loss (late loss or no late loss).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Arm (Active Comparator): Open-label low-molecular-weight heparin (LMWH) prophylaxis until 37 weeks gestation AND low-dose aspirin daily until delivery.
  Interventions: Drug: Low-molecular-weight heparin
- Experimental Arm (Experimental): Open-label low-dose Aspirin 81 mg daily from randomization until delivery.
  Interventions: Drug: Aspirin 81 mg

INTERVENTIONS:
Drug: Aspirin 81 mg — Aspirin 81 mg po daily in tablet form.
  Other Names: Acetylsalicylic Acid
  Arms: Experimental Arm
Drug: Low-molecular-weight heparin — The LMWH regime will be at the discretion of the treating physician, with a suggested regime as follows: tinzaparin 4,500 IU sc daily until 20 weeks gestation, and then 4,500 IU sc twice daily until 37 weeks gestation.
  Other Names: Tinzaparin; Dalteparin; Enoxaparin; LMWH
  Arms: Standard of Care Arm

SUMMARY:
The APPLE pilot trial is a feasibility study that is a multicentre, open-label, randomized controlled trial. Pregnant women with antiphospholipid syndrome (APS) and a history of late (≥10 weeks gestation) or recurrent early (2 <10 weeks) pregnancy loss will be recruited.

Eligible and consenting subjects will be assigned to one of two study arms: open-label low-molecular-weight heparin (LMWH) prophylaxis until 37 weeks gestation AND low-dose aspirin (ASA) daily until delivery, or open-label low-dose aspirin daily from randomization until delivery.

DETAILED DESCRIPTION:
The purpose of this pilot trial is to determine the feasibility of conducting a multicenter randomized full trial evaluating antepartum prophylaxis with ASA versus LMWH/ASA in women with confirmed APS and a history of late or recurrent early pregnancy loss.

Given the large sample size needed to adequately power a large multicenter trial that assesses the efficacy of ASA alone versus LMWH/ASA, the investigators first need to determine if it is possible to meet minimum recruitment rates needed for a full multicenter trial. If the pilot feasibility trial is successful, then the secondary outcomes collected will be used in the analysis of the full multicenter trial.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pregnancy;
* 18 years or older;
* Two or more unexplained pregnancy loss before the 10th week of gestation, AND/OR one or more unexplained pregnancy loss at or beyond the 10th week of gestation;
* One or more APS laboratory criteria present, according to the revised Sapporo criteria;

Exclusion Criteria:

* Greater than 11 weeks +6 days gestational age at time of randomization;
* Indication(s) for prophylactic or therapeutic-dose anticoagulation;
* Contraindication to heparin or aspirin;
* Received 7 or more doses of LMWH;
* Previous participation in the trial;
* Geographic inaccessibility;
* Refused consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Rodger, MD, Principal Investigator — Ottawa Hospital Research Institute; Leslie Skeith, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamulyak EN, Scheres LJ, Marijnen MC, Goddijn M, Middeldorp S. Aspirin or heparin or both for improving pregnancy outcomes in women with persistent antiphospholipid antibodies and recurrent pregnancy loss. Cochrane Database Syst Rev. 2020 May 2;5(5):CD012852. doi: 10.1002/14651858.CD012852.pub2. PMID 32358837

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care Arm | Experimental Arm
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 0 participants were enrolled in the standard of care arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Arm | Experimental Arm | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Study Feasibility: Mean Recruitment Rate Per Center Per Month
Description: The primary feasibility outcome of the pilot trial is the mean recruitment rate per center per month.
Time Frame: 24 months
Population: 1 participant was recruited (ASA alone arm) and the pilot trial was stopped early due to feasibility.
Measure: Number; unit: participants
Arm/Group | Standard of Care Arm | Experimental Arm
Number analyzed (Participants) | 0 | 1
participants |  | 1

2. Secondary Outcome: Essential Documents
Description: Proportion of sites requiring >18 months to obtain all required approvals/contracts from time of delivery of all study documents.
Time Frame: 18 months
Population: Site #1 was able to obtain all applicable approvals and begin recruitment in 12 months. Not applicable applicable for site #2 as study was closed early due to low recruitment.
Measure: Number; unit: Sites
Groups:
- Approval Timeline: Sites requiring >18 months for all approvals
Arm/Group | Approval Timeline
Number analyzed (Participants) | 1
Sites | 1

3. Secondary Outcome: Eligibility
Description: Proportion of screened patients who meet eligibility criteria (i.e. patients who meet inclusion criteria and are also eligible based on exclusion criteria).
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Screened Patients Who Met Eligibility Criteria: Screened patients who meet eligibility criteria
Arm/Group | Screened Patients Who Met Eligibility Criteria
Number analyzed (Participants) | 25
Participants | 4

4. Secondary Outcome: Consent
Description: Proportion of eligible subjects who provide consent.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Consented Eligible Patients: Eligible patients who provided consent
Arm/Group | Consented Eligible Patients
Number analyzed (Participants) | 4
Participants | 1

5. Secondary Outcome: Withdrawals/Loss to Follow-up
Description: Proportion of withdrawals/loss to follow-up among randomized patients.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Withdrawal/Lost to Follow-up: Withdrawal/Lost to follow-up among randomized patients
Arm/Group | Withdrawal/Lost to Follow-up
Number analyzed (Participants) | 1
Participants | 0

6. Secondary Outcome: Crossover Rate
Description: Crossover rate between standard of care and experimental study arms.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Crossover Rate: Crossover rate between standard of care and experimental study arms.
Arm/Group | Crossover Rate
Number analyzed (Participants) | 1
Participants | 0

7. Secondary Outcome: Study Drug Compliance
Description: Level of compliance with study drug through patient recall and patient medication diary.
Time Frame: 52 weeks
Population: No participants in standard of care arm
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Experimental Arm
Number analyzed (Participants) | 0 | 1
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: The AE reporting period for this trial begun upon randomization, and ended 30 days after receiving the last dose of study drug.
Description: AEs were elicited, monitored and recorded throughout the study. For each participant, AEs were submitted to the trial office after each follow-up visit. The investigator is to report all directly observed AEs and all AEs spontaneously reported by the participant. In addition, each participant will be questioned about AEs at each clinic visit following initiation of treatment.
Arm/Group | Standard of Care Arm | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT03100123/Prot_SAP_000.pdf